CLINICAL TRIAL: NCT06719739
Title: Clinical Outcomes in Cataract Patients with Macular Epiretinal Membrane After Implantation of Functional Intraocular Lenses
Brief Title: Functional IOL Implantation in Patients with Epiretinal Membrane
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jin Yang, Professor, Eye & ENT Hospital of Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Mild ERM and IOL Implantation
Record Dates: First submitted 2024-12-04; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cataract; Intraocular Lens Complication; Epiretinal Membrane
MeSH Terms: conditions — Cataract; Epiretinal Membrane | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Functional IOL (Experimental): Experimental group
  Interventions: Device: Intraocular lens implantation
- Monofocal IOL (Other): Control Group
  Interventions: Device: Intraocular lens implantation

INTERVENTIONS:
Device: Intraocular lens implantation — Cataract patients scheduled for surgery will be evaluated by OCT, and those diagnosed with macular epiretinal membrane will be implanted in different IOLs according to the patients' decision: monodical IOL or functional IOL.

SUMMARY:
We have designed this prospective study to evaluate macular involvement and epiretinal membrane (ERM) grading by OCT in eyes with ERM and to compare clinical outcomes after implantation of Enhance IOL with standard monofocal IOL in eyes with ERM grading preoperatively, aiming to find out whether functional IOL is benefit for patients with ERM.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, comparative study. Cataract patients scheduled for surgery will be evaluated by OCT, and those diagnosed with grade-1 macular epiretinal membrane will be implanted in different IOLs according to the patients' decision: monofocal IOL or functional IOL. The follow-up duration sets to be 2-years. Outcome measures: The primary outcome measure is visual acuity measured according to UDVA and CDVA at 5 m; UIVA at 66 cm; and UNVA at 40 cm. Visual examination will be performed twice under sufficient lighting, and the international standard visual acuity table will be used. The secondary outcome measures are as follows: (1) OCT examination and Amsler grid test. (2) HOA such as coma, spherical, trefoil, and secondary astigmatism will be measured using internal and total values at a 3-mm pupil size with the HOYA iTrace ray-tracing system (Tracey Technologies, Houston, TX, USA); (3) Modulation transfer function (MTF) curve and Strehl ratio (SR) will be also measured using internal and total values at a 3-mm pupil size with the HOYA iTrace ray-tracing system; (4) Defocus curves for each IOL will be obtained by plotting the mean visual acuity with 13 values of defocus from +2.0 D to -4.0 D on the ETDRS chart in logMAR units. The defocus curve simulates the patient's visual acuity at different distances by placing positive and negative lenses in 0.5 D increments in front of the patient's eyes. The measurements will be performed by adding lenses to CDVA; (5) Contrast sensitivity (CS) will be assessed with best distance correction using the Optec6500 (Stereo Optical Co., Inc., Chicago, IL, USA). Assessments will be made at spatial frequencies of 1.5, 3, 6, 12, and 18 cycles per degree (cpd), with or without glare, under photopic or mesopic conditions (background luminance of 85 cd/m2 or 3 cd/m2). CS value refers to the value of the last patch that can be recognized, and all patients will see at least one patch. All CS data will be transformed to logarithmic units and log CS values for analysis; (6) Reading ability will be measured by the Chinese Reading Visual Acuity Chart (CRVAC) at near and intermediate distances. With the CRVAC, reading acuity (in logMAR) and reading speed (in words per minute) can be measured at a predetermined or preferred distance successively. The minimum distinguishable font size and corresponding visual acuity of the patients with UNVA and UIVA above 0.1 LogMAR will be respectively measured at 66 cm and 40 cm under photopic conditions. The patients will be required to read a text with a font size of 5 point (LogMAR 0.5) at 40cm and of 8 point (LogMAR 0.7) at 66cm. The reading time will be timed and converted to words per minute; and (7) the functional vision and incidence of photic phenomena will be surveyed using VF-14 questionnaire and Qov questionnaire which are attached in the supplementary materials. Study population >90 subjects/ 90 eyes (45 eyes per group, total 2 groups) Primary/Secondary endpoints (or perhaps exploratory endpoint) The primary endpoint of this study is to demonstrate the noninferiority of functional IOL group to monodical IOL group in mean CDVA and UDVA (5m) postoperatively. If the primary endpoint is met, the first secondary endpoint is to demonstrate superiority of ICB00 group to DCB00 group in mean UIVA (66cm) and UNVA (40cm). The prespecified Snellen equivalent targets of ICB00 group are determined and included the following: 20/25 or better photopic UIVA (measured at 66 cm); 20/40 (0.5 decimal) or better photopic UNVA at 40 cm. Additional secondary endpoints are to compare the defocus curve behaviour, objective visual quality, reading ability and subject satisfaction between the two groups. Study Timeline Visit Schedule

1.Baseline visit 2.2. 1-day visit 3.3. 1-week visit 4.4. 1-month visit 5.5. 3-month visit 6.6. 6-month visit 7.7. 1-year visit 8.8. 2-year visit

ELIGIBILITY:
Inclusion Criteria:

* Requirement for cataract extraction
* Age > 40 years
* Axial length in 21mm to 25mm
* ERM

Exclusion Criteria:

* Residual corneal astigmatism > 1.0 D
* Amblyopia
* Previous ocular surgery
* Other ocular pathologies apart from mERM, such as diabetic retinopathy, macular degeneration, glaucoma with field defects
* Requirements for further ocular surgery (other than Nd:YAG capsulotomy) or retinal laser treatments during the study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
UDVA | 1-day/1-week/1-month/3-months/6-monhts/1-year/2-years
  Uncorrected distance visual acuity

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Eye and Ear, Nose, and Throat Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Heping Eye Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No